CLINICAL TRIAL: NCT06259630
Title: Effect of Nicotine on Acquisition and Extinction of a Conditioned Place Preference in a Virtual Reality Environment
Brief Title: Nicotine Virtual Reality Conditioned Place Preference
Acronym: NEVE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigators no longer wanted to pursue this research topic
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB15-1337
Record Dates: First submitted 2017-02-15; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Nicotine Addiction; Nicotine Use Disorder
Keywords: Nicotine
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo followed by Nicotine Arm (Experimental): Participant receives placebo on day 1 and nicotine on day 2.
  Interventions: Drug: Nicotine; Drug: Placebo oral capsule
- Nicotine followed by Placebo Arm (Experimental): Participant receives nicotine on day 1 and placebo on day 2.
  Interventions: Drug: Nicotine; Drug: Placebo oral capsule
- Placebo followed by Placebo Arm (Placebo Comparator): Participant receives placebo on day 1 and day 2.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Nicotine — Participant receives oral dose of nicotine
  Arms: Nicotine followed by Placebo Arm; Placebo followed by Nicotine Arm
Drug: Placebo oral capsule — Participant receives oral dose of placebo

SUMMARY:
In this between-subjects, placebo controlled, double-blind study, the investigators will examine the effects of low oral doses of nicotine on the learning and extinction of a conditioned place preference acquired in a virtual reality environment by healthy human subjects. Physiological and subjective responses to the drug will also be monitored.

DETAILED DESCRIPTION:
External cues and contexts contribute to the development of smoking and the use of other drugs, and drugs themselves can alter the value of conditioned cues. Interestingly, nicotine increases the acquisition of new learning, and has been considered as a "cognitive enhancer". Nicotine also prolongs responding when responding is no longer rewarded, during extinction. Although many studies have examined the effects of drugs on learning (acquisition) and unlearning (extinction) in laboratory animals, few have investigated drug effects on learning in humans. Recently, novel procedures have been developed to study conditioning in humans, pairing initially neutral places with food, money or drugs. The investigators will use one of these procedures, a virtual place conditioning procedure, to study how nicotine affects the acquisition and extinction of conditioned behaviors in humans.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have at least a high school education and be in good physical and mental health.

Exclusion Criteria:

* Individuals with current medical conditions, and/or a history of serious medical problems (e.g., cardiac, kidney, liver, and neurological).

Additional Exclusion Criteria include:

* regular medication,
* pregnancy,
* color blindness,
* left-handedness,
* consumption of 5 or more cigarettes per day,
* English non-fluency and current DSM-IV Axis 1 diagnosis excluding nicotine dependence.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Virtual Environment "Liking" | Participant rate on a visual analog scale how much they prefer one virtual environment over another

SECONDARY OUTCOMES:
Time spent in virtual environment | Participants actively choose which environment to spend time in. The length of those virtual visits is measured and compared during the study sessions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center - Human Behavioral Pharmacology Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acheson A, Mahler SV, Chi H, de Wit H. Differential effects of nicotine on alcohol consumption in men and women. Psychopharmacology (Berl). 2006 May;186(1):54-63. doi: 10.1007/s00213-006-0338-y. Epub 2006 Mar 25. PMID 16565827
- [Background] Astur RS, Carew AW, Deaton BE. Conditioned place preferences in humans using virtual reality. Behav Brain Res. 2014 Jul 1;267:173-7. doi: 10.1016/j.bbr.2014.03.018. Epub 2014 Mar 20. PMID 24657735
- [Background] Caggiula AR, Donny EC, White AR, Chaudhri N, Booth S, Gharib MA, Hoffman A, Perkins KA, Sved AF. Environmental stimuli promote the acquisition of nicotine self-administration in rats. Psychopharmacology (Berl). 2002 Sep;163(2):230-7. doi: 10.1007/s00213-002-1156-5. Epub 2002 Jul 13. PMID 12202970
- [Background] Childs E, de Wit H. Amphetamine-induced place preference in humans. Biol Psychiatry. 2009 May 15;65(10):900-4. doi: 10.1016/j.biopsych.2008.11.016. Epub 2008 Dec 25. PMID 19111278
- [Background] Everitt BJ. Neural and psychological mechanisms underlying compulsive drug seeking habits and drug memories--indications for novel treatments of addiction. Eur J Neurosci. 2014 Jul;40(1):2163-82. doi: 10.1111/ejn.12644. Epub 2014 Jun 17. PMID 24935353
- [Background] Guy EG, Fletcher PJ. The effects of nicotine exposure during Pavlovian conditioning in rats on several measures of incentive motivation for a conditioned stimulus paired with water. Psychopharmacology (Berl). 2014 Jun;231(11):2261-71. doi: 10.1007/s00213-013-3375-3. Epub 2013 Dec 7. PMID 24317443
- [Background] Hukkanen J, Jacob P 3rd, Benowitz NL. Metabolism and disposition kinetics of nicotine. Pharmacol Rev. 2005 Mar;57(1):79-115. doi: 10.1124/pr.57.1.3. PMID 15734728
- [Background] Hutton-Bedbrook K, McNally GP. The promises and pitfalls of retrieval-extinction procedures in preventing relapse to drug seeking. Front Psychiatry. 2013 Mar 12;4:14. doi: 10.3389/fpsyt.2013.00014. eCollection 2013. PMID 23487003
- [Background] Molet M, Billiet G, Bardo MT. Conditioned place preference and aversion for music in a virtual reality environment. Behav Processes. 2013 Jan;92:31-5. doi: 10.1016/j.beproc.2012.10.001. Epub 2012 Oct 23. PMID 23089383
- [Background] Tian S, Gao J, Han L, Fu J, Li C, Li Z. Prior chronic nicotine impairs cued fear extinction but enhances contextual fear conditioning in rats. Neuroscience. 2008 Jun 2;153(4):935-43. doi: 10.1016/j.neuroscience.2008.03.005. Epub 2008 Mar 8. PMID 18440720
- [Background] Tzschentke TM. Measuring reward with the conditioned place preference paradigm: a comprehensive review of drug effects, recent progress and new issues. Prog Neurobiol. 1998 Dec;56(6):613-72. doi: 10.1016/s0301-0082(98)00060-4. PMID 9871940
- [Background] Wignall ND, de Wit H. Effects of nicotine on attention and inhibitory control in healthy nonsmokers. Exp Clin Psychopharmacol. 2011 Jun;19(3):183-91. doi: 10.1037/a0023292. PMID 21480731
- [Background] Gould TJ, Collins AC, Wehner JM. Nicotine enhances latent inhibition and ameliorates ethanol-induced deficits in latent inhibition. Nicotine Tob Res. 2001 Feb;3(1):17-24. doi: 10.1080/14622200020032060. PMID 11260807
- [Background] Fond G, Micoulaud-Franchi JA, Brunel L, Macgregor A, Miot S, Lopez R, Richieri R, Abbar M, Lancon C, Repantis D. Innovative mechanisms of action for pharmaceutical cognitive enhancement: A systematic review. Psychiatry Res. 2015 Sep 30;229(1-2):12-20. doi: 10.1016/j.psychres.2015.07.006. Epub 2015 Jul 8. PMID 26187342
- [Background] Chaudhri N, Caggiula AR, Donny EC, Booth S, Gharib M, Craven L, Palmatier MI, Liu X, Sved AF. Operant responding for conditioned and unconditioned reinforcers in rats is differentially enhanced by the primary reinforcing and reinforcement-enhancing effects of nicotine. Psychopharmacology (Berl). 2006 Nov;189(1):27-36. doi: 10.1007/s00213-006-0522-0. Epub 2006 Sep 22. PMID 17019569
- [Background] Folstein MF, Luria R. Reliability, validity, and clinical application of the Visual Analogue Mood Scale. Psychol Med. 1973 Nov;3(4):479-86. doi: 10.1017/s0033291700054283. No abstract available. PMID 4762224
- [Background] Adam KC, Mance I, Fukuda K, Vogel EK. The contribution of attentional lapses to individual differences in visual working memory capacity. J Cogn Neurosci. 2015 Aug;27(8):1601-16. doi: 10.1162/jocn_a_00811. Epub 2015 Mar 26. PMID 25811710